CLINICAL TRIAL: NCT02699996
Title: Promoting Follow-Up Care Self-Management for Adolescent and Young Adult (AYA) Childhood Cancer Survivors
Brief Title: Peer Mentoring in Promoting Follow-up Care Self-Management in Younger Childhood Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katie Devine, PhD, MPH, Assistant Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro20150001955; NCI-2015-02098 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20150001955; 131507 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2016-03-01; First posted 2016-03-07 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Cancer Survivor
Keywords: Cancer Survivor; Young Adult; Peer Mentor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- self-management + peer mentoring (Experimental): Participants complete the self-management + peer mentoring intervention comprising 5 online educational modules and 6 videoconference or phone calls with the peer mentor.
  Interventions: Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Questionnaire Administration — Complete interview
Behavioral: Telephone-Based Intervention — Complete the self management + peer mentoring intervention with videoconferencing

SUMMARY:
This pilot trial studies a peer mentoring and online self-management program to see how well it works in promoting follow-up care self-management in younger childhood cancer survivors. Childhood cancer survivors require lifelong follow-up care to identify, monitor, and treat medical and psychosocial late effects stemming from their cancer, its treatment, and lifestyle factors. A peer mentoring program + self-management may improve disease knowledge, health motivation, problem-solving skills, stress management, and communication with caregivers and providers in adolescent and young adult cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility of the self-management + peer mentoring program in a pilot trial.

II. Assess preliminary outcomes of the peer mentoring program.

OUTLINE:

All Participants will be asked to complete online self-management educational modules and 6 weekly peer mentor calls to facilitate engagement with the online modules and offer specialized support. We will also recruit and train peer Mentors.

ELIGIBILITY:
Inclusion Criteria:

PEER MENTOR ELIGIBILITY:

* Age 21-29
* At least 1.5 years from treatment
* Self-reported primary responsibility for care and "complete readiness" using the Readiness for Transition Questionnaire

PATIENT ELIGIBILITY:

* Age 18-25
* At least 1.5 years from treatment
* Currently does not independently self-manage follow-up care according to self-report to assume total responsibility for care (i.e., reports low readiness [score of 1 or 2 out of 4] OR scores <3 on any of the 10-item responsibility scale from the Readiness for Transition Questionnaire)

Exclusion Criteria:

PATIENT EXCLUSION CRITERIA: Physician- or self-reported cognitive delay or impairment that would prevent self-management of healthcare

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Devine, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Intervention Participants; Group Intervention Mentors: one arm, all participants complete 6 week self-management (5 online educational modules) + peer mentoring (6 video-conference or phone calls) intervention.
Period: Overall Study
Arm/Group | Group Intervention Participants | Group Intervention Mentors
Started | 20 | 11
Completed | 15 | 9
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Population: Group Intervention Participants: all completed baseline survey. Group Intervention Mentors: all completed Mentor training.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Intervention Participants | Group Intervention Mentors | Total
Number analyzed (Participants) | 20 | 11 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 11 | 31
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 11 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 17 | 10 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Study Enrollment Rates, Retention Rates, Adherence to the Intervention, and Reasons for Study Drop Out.
Description: Descriptive analyses will be used to evaluate expected enrollment (> 50%), retention (> 80%), and completion of intervention sessions (> 75%).
Time Frame: 6 weeks
Population: Group Intervention Participants: the total number of potential participants identified by the Cancer Registry, whose contact information was provided to our study team for recruitment. Group Intervention Mentors-identified and recommended by the local survivorship clinic physicians and clinical staff.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Intervention Participants | Group Intervention Mentors
Number analyzed (Participants) | 36 | 11
Participants
  Study Enrollment Rates: Eligible on study | 20 | 11
  Study Enrollment Rates: Ineligible | 8 | 0
  Study Enrollment Rates: Declined participation/No time | 1 | 0
  Study Enrollment Rates: Unable to reach | 7 | 0
  Reason Study Drop Out: number analyzed (Participants) | 5 | 2
  Reason Study Drop Out: Eligible on study | 0 | 0
  Reason Study Drop Out: Ineligible | 0 | 0
  Reason Study Drop Out: Declined participation/No time | 1 | 2
  Reason Study Drop Out: Unable to reach | 4 | 0
  Participant Retention Rates: number analyzed (Participants) | 20 | 11
  Participant Retention Rates: Eligible on study | 15 | 9
  Participant Retention Rates: Ineligible | 0 | 0
  Participant Retention Rates: Declined participation/No time | 1 | 2
  Participant Retention Rates: Unable to reach | 4 | 0
  Adherence to Sessions: number analyzed (Participants) | 15 | 9
  Adherence to Sessions: Eligible on study | 15 | 9
  Adherence to Sessions: Ineligible | 0 | 0
  Adherence to Sessions: Declined participation/No time | 0 | 0
  Adherence to Sessions: Unable to reach | 0 | 0

2. Primary Outcome: Satisfaction With Intervention, Measured by 1) General Satisfaction, 2) Intervention Utility Questionnaire, 3) Impact Questionnaire (i.e., Effectiveness), and 4) Adherence Questionnaire ( i.e., Barriers to Engagement).
Description: 1. General Satisfaction: Average of each item reported separately. 1: Program; 2: Online educational materials; 3: Discussion with mentor; 4: Frequency of calls; 5: Program duration; 6: Material read. Items 1, 2, 3, & 6 are rated on a 1 "not at all" to 5 "very" scale (higher=higher satisfaction). Item 4 uses a 1 "not frequent enough" to 3 "too frequent" scale. Item 5 uses a 1 "way too short" to 5 "way too long" scale.
  2. 12-items adapted from Internet Intervention Utility Questionnaire; measures perceived usefulness on 1 "not at all" to 5 "very" scale, higher=higher usefulness. Average total score reported.
  3. 16-item Impact Questionnaire measures perceived effectiveness in improving targeted skills using 1 "not at all" to 5 "very" scale (higher=greater perceived effectiveness). Average total score reported.
  4. 6-item Adherence Questionnaire measures barriers to engagement using 1 "not a problem" to 3 "major problem" scale. (higher=bigger barrier). Average total score reported.
Time Frame: 6 weeks (post-intervention)
Population: Satisfaction with intervention, administered to all Participants, i.e., Group Intervention Participants, n=15.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Intervention Participants
Number analyzed (Participants) | 15
score on a scale
  Satisfaction w/Program [Range 1-5] | 4.20 (0.86)
  Satisfaction w/Online materials [Range 1-5] | 3.80 (1.01)
  Satisfaction w/Discussions [Range 1-5] | 4.60 (0.63)
  Frequency of calls [Range 1-3; 2="Just right"] | 2.0 (0.39)
  Program duration [Range 1-5;3="Just right"] | 3.07 (0.59)
  Amount of ed materials read [Range 1-5] | 3.80 (1.01)
  Internet Utility Total Score [Range 1-5] | 3.96 (0.69)
  Impact Questionnaire Total Score [Range 1-5] | 3.81 (0.90)
  Adherence Questionnaire Total [Range 1-3] | 1.12 (0.21)

3. Primary Outcome: Mentor Training Satisfaction
Description: Mentor 6-item Training Satisfaction measured on a scale from 1 "strongly disagree" to 4 "strongly agree" (higher score=high satisfaction). Administered to Group Intervention Mentors only. Total average score is reported.
Time Frame: Time of enrollment, after completing mentor training.
Population: Mentors completed satisfaction with training questionnaire after completion of the Mentor Training and prior to being matched with a participant (mentee).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Intervention Mentors
Number analyzed (Participants) | 11
score on a scale | 3.92 (0.16)

4. Secondary Outcome: Transition Readiness, as Measured by the Readiness for Transition Questionnaire - Survivor Version
Description: Respondents rate how responsible they are for various healthcare tasks on a 4-point scale, where 1= "not responsible at all", and 4= "almost always responsible." The Adolescent Responsibility Scale is calculated by averaging responses across all 10 items (RTQ-Survivor). A single item assessing "overall readiness to assume complete responsibility for health care" on the same 4-point scale is analyzed separately.
Time Frame: Baseline to up to 6 weeks
Population: All participants who completed baseline assessment, intervention, and follow-up assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Intervention Participants
Number analyzed (Participants) | 15
score on a scale
  RTQ-Survivor Adolescent Responsibility pre- | 3.08 (0.69)
  RTQ-Survivor Adolescent Responsibility post- | 3.60 (0.35)
  RTQ-Overall Readiness pre- | 2.60 (0.74)
  RTQ-Overall Readiness post- | 3.27 (0.70)
Statistical Analysis 1: Comparison: Group Intervention Participants; RTQ-Survivor Adolescent Responsibility Score; Test type: Superiority; p < .01, t-test, 2 sided; df = 14; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [0.17 to 0.86]
Statistical Analysis 2: Comparison: Group Intervention Participants; RTQ-Overall Readiness Score; Test type: Superiority; p < .01, t-test, 2 sided; df=14; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [0.27 to 1.07]

5. Secondary Outcome: Transition Readiness, as Measured by the Transition Readiness Inventory (Phase 2).
Description: The Transition Readiness Inventory (TRI) yields six sub-scale scores: Knowledge, Skills/Self-Efficacy, Beliefs/Expectations, Goals/Motivation, Relationship/Communication, and Psychosocial/Emotional. Total average score is reported across all sub-scales (TRI-total), as well as each sub-scale total score. Scores are averaged across items on a 5-point scale from 1 "not at all" to 5 "extremely" or "always," with higher scores indicating better functioning.
Time Frame: Baseline to up to 6 weeks
Population: Participants who completed baseline, intervention, and follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Intervention Participants
Number analyzed (Participants) | 15
score on a scale
  TRI-total pre- | 4.03 (0.41)
  TRI-total post- | 4.27 (0.23)
  TRI Knowledge pre- | 4.21 (0.63)
  TRI Knowledge post- | 4.70 (0.37)
  TRI Skills/Self-Efficacy pre- | 3.97 (0.65)
  TRI Skills/Self-Efficacy post- | 4.27 (0.47)
  TRI Beliefs/Expectations pre- | 3.93 (0.39)
  TRI Beliefs/Expectations post- | 4.06 (0.34)
  TRI Goals/Motivation pre- | 4.15 (0.77)
  TRI Goals/Motivation post- | 4.55 (0.54)
  TRI Relationship/Communication pre- | 4.23 (0.40)
  TRI Relationship/Communication post- | 4.28 (0.40)
  TRI Psychosocial/Emotional pre- | 3.69 (0.73)
  TRI Psychosocial/Emotional post- | 3.79 (0.40)
Statistical Analysis 1: Comparison: Group Intervention Participants; TRI-total Score; Test type: Superiority; p = 0.02, t-test, 2 sided; df=14; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [0.05 to 0.42]
Statistical Analysis 2: Comparison: Group Intervention Participants; TRI Knowledge score; Test type: Superiority; p < .01, t-test, 2 sided; df=14; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [0.26 to 0.73]
Statistical Analysis 3: Comparison: Group Intervention Participants; TRI Skills/Self-Efficacy Score; Test type: Superiority; p = 0.053, t-test, 2 sided; df=14; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.0044 to 0.60]
Statistical Analysis 4: Comparison: Group Intervention Participants; TRI Beliefs/Expectations score; Test type: Superiority; p = 0.03, t-test, 2 sided; df=14; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [0.02 to 0.24]
Statistical Analysis 5: Comparison: Group Intervention Participants; TRI Goals/Motivation score; Test type: Superiority; p < .01, t-test, 2 sided; df=14; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [0.11 to 0.69]
Statistical Analysis 6: Comparison: Group Intervention Participants; Relationship/Communication Score; Test type: Superiority; p = 0.61, t-test, 2 sided; df=14; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.16 to 0.26]
Statistical Analysis 7: Comparison: Group Intervention Participants; TRI Psychosocial/Emotional Score; Test type: Superiority; p = 0.65, t-test, 2 sided; df=14; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.37 to 0.57]

6. Secondary Outcome: Symptoms of Depression, as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short-Form (v1.0 8b).
Description: Respondents report symptoms on a 5-point rating scale from 1 "never" to 5 "always" in the past 7 days, with higher scores indicating higher levels of negative affect. A total raw summary score is calculated and then translated into a standardized T-score with a mean of 50 and standard deviation of 10.
Time Frame: Baseline to up to 6 weeks
Population: We had missing data for one participant, therefore total number of participants analyzed is 14.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Group Intervention Participants
Number analyzed (Participants) | 14
T-score
  Depression pre- | 52.66 (12.15)
  Depression post- | 51.02 (9.63)
Statistical Analysis 1: Comparison: Group Intervention Participants; Test type: Superiority; p = .56, t-test, 2 sided; df = 13; Median Difference (Final Values) = -1.64, 95% CI 2-sided [-7.62 to 4.34]

7. Secondary Outcome: Symptoms of Anxiety, as Measured by the PROMIS Anxiety Short-Form (v1.0 8a)
Description: as for outcome 6
Time Frame: Baseline to up to 6 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Group Intervention Participants
Number analyzed (Participants) | 15
T-score
  Anxiety pre- | 59.29 (14.20)
  Anxiety post- | 57.55 (7.97)
Statistical Analysis 1: Comparison: Group Intervention Participants; Test type: Superiority; p = .42, t-test, 2 sided; df = 14; Mean Difference (Final Values) = -1.74, 95% CI 2-sided [-6.23 to 2.75]

8. Secondary Outcome: Cancer Related Worry Scale
Description: This 4-item scale is measuring cancer-related worries (i.e., recurrence of cancer, future diagnostic tests, cancer coming back, other type of cancer). A total score is calculated by averaging across items on a 5-point scale (from 1="Strongly disagree" to 5="Strongly agree"), with higher scores indicating greater worry. Total average score is reported.
Time Frame: Baseline to up to 6 weeks
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Intervention Participants
Number analyzed (Participants) | 15
score on a scale
  Cancer Related Worry pre- | 3.72 (1.20)
  Cancer Related Worry post- | 3.43 (1.41)
Statistical Analysis 1: Comparison: Group Intervention Participants; Test type: Superiority; p = .26, t-test, 2 sided; df = 14; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.80 to 0.23]

9. Secondary Outcome: Short Grit Scale
Description: Perseverance is measured via the The Short Grit Scale, an 8-item measure of perseverance for long-term goals. A total scale score is calculated by averaging across all items, on a 5-point scale (from 1 "not at all like me" to 5 "very much like me"), with higher scores indicating greater perseverance.
Time Frame: Baseline to up to 6 weeks
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Intervention Participants
Number analyzed (Participants) | 15
score on a scale
  Grit pre- | 3.29 (0.63)
  Grit post- | 3.57 (0.58)
Statistical Analysis 1: Comparison: Group Intervention Participants; Test type: Superiority; p = .03, t-test, 2 sided; df = 14; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [0.03 to 0.52]

10. Secondary Outcome: Impact of Cancer, as Measured by Three Subscales of the Impact of Cancer - Childhood Cancer Survivors Scale
Description: The three subscales measure perceptions of cancer impact on Body Health (8 items), Personal Growth (5 items), and Memory Problems (4 items). Sub-scales are scored by averaging across items using a 5-point scale (where 1="not at all", and 5="very much"), with higher scores indicating greater impact.
Time Frame: Baseline to up to 6 weeks
Population: Participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Intervention Participants
Number analyzed (Participants) | 15
score on a scale
  Body Health pre- | 3.60 (1.13)
  Body Health post- | 3.80 (0.86)
  Personal Growth pre- | 4.39 (0.67)
  Personal Growth post- | 4.25 (0.58)
  Memory pre- | 3.02 (0.43)
  Memory post- | 3.12 (0.56)
Statistical Analysis 1: Comparison: Group Intervention Participants; Body Health Subscale; Test type: Superiority; p = .20, t-test, 2 sided; df = 14; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.12 to 0.52]
Statistical Analysis 2: Comparison: Group Intervention Participants; Personal Growth Subscale; Test type: Superiority; p = .40, t-test, 2 sided; df = 14; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.46 to 0.20]
Statistical Analysis 3: Comparison: Group Intervention Participants; Memory Subscale; Test type: Superiority; p = .29, t-test, 2 sided; df = 14; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.09 to 0.29]

11. Secondary Outcome: Barriers to Follow-up Care & Adherence
Description: Barriers to follow-up care & adherence evaluated by insurance status, current provider, and other barriers to care using 6 items from the Follow-Up Care Use and Health Outcomes of Cancer Survivors (FOCUS). Participants report on appointments, cancer screening, and other adherence markers on a 5-point scale (from 1="Strongly disagree" to 5="Strongly agree"), where higher score indicates grater barrier. Total average score is reported.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Intervention Participants
Number analyzed (Participants) | 15
score on a scale
  Barriers pre- | 2.20 (0.47)
  Barriers post- | 2.01 (0.59)
Statistical Analysis 1: Comparison: Group Intervention Participants; Test type: Superiority; p = .08, t-test, 2 sided; df = 14; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.40 to 0.03]

ADVERSE EVENTS:
Time Frame: For the study duration, i.e., ~6 weeks for each participant.
Arm/Group | Group Intervention Participants | Group Intervention Mentors
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/11
Other Adverse Events (participants affected / at risk) | 0/20 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT02699996/Prot_SAP_000.pdf